CLINICAL TRIAL: NCT06182514
Title: State of Play at the SAMU 67: What Are the Themes Mainly Concerned by the Second Intention SMUR, Called Reinforcements, on the Sector of the Bas-Rhin? Are There Modifiable Factors That Could Allow us to Anticipate Them Better
Brief Title: What Are the Main Themes Concerned by the Second-line SMUR 67, Known as Reinforcements, in the Bas-Rhin Sector
Acronym: RenforSMUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8675
Record Dates: First submitted 2022-09-06; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Reasons for Emergency Calls
Keywords: emergency calls; SAMU67; SMUR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators wish to evaluate the possibility of anticipating the requests for SMUR reinforcement within the SAMU67.

The studied population concerns each patient having benefited from an SMUR at the time of his pre-hospital care. The investigators expect from this study an improvement of the assumption of responsibility of the patients in the future with optimization of the delay of sending of an SMUR when this one is necessary.

ELIGIBILITY:
Inclusion criteria:

* Adult patients having benefited from a pre-hospital SMUR over the period from 01/01/2020 to 14/07/2020.
* No opposition from the patient or his parental authority to the re-use of his medical data for scientific research.

Exclusion criteria:

- Presence of opposition from the patient or his parental authority to the re-use of his medical data for scientific research purposes.

Min Age: 1 Month | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients having benefited from a pre-hospital SMUR over the period from 01/01/2020 to 14/07/2020.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the main reasons and themes of patient calls leading to the Emergency Medical Service being sent for reinforcement | Through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urgences Médico-Chirurgicales Adules, Strasbourg, France